CLINICAL TRIAL: NCT00355680
Title: Comparative Study of Indigenous Green Laser With Already Available Green Laser in Proliferative Diabetic Retinopathy
Brief Title: Green Laser Photocoagulation Study in Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aurolab (Other)
Collaborators: Raja Ramanna Centre for Advanced Technology (RRCAT) (Unknown)
Responsible Party: A. Heber, Aurolab
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2PR1210511
Record Dates: First submitted 2006-07-21; First posted 2006-07-24 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Diabetic Retinopathy
Keywords: Retina; Retinal Diseases; Retinal Vessels; Laser Coagulation
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Aurolab Green Laser
  Interventions: Device: Green Laser (Aurolas, Aurolab)
- 2 (Active Comparator): Available Green Laser
  Interventions: Device: Green Laser (Iridex)

INTERVENTIONS:
Device: Green Laser (Aurolas, Aurolab) — Green laser developed by Aurolab
  Other Names: Aurolas
  Arms: 1
Device: Green Laser (Iridex) — Already available green laser
  Other Names: Iridex
  Arms: 2

SUMMARY:
To Demonstrate that indigenous green laser produces similar treatment effect on the retina when compared with already available green laser.

DETAILED DESCRIPTION:
Proliferative Diabetic Retinopathy is ocular pathology in poor glycaemic controlled Diabetic patient Characterized by micro-vascular pathology with capillary closure in the retina leading to hypoxia of tissue there by formation of immature vessels to provide better oxygenation of retinal tissue.

In this randomized double blinded study a convenient sample size of 24 eyes assigned to compare indigenously developed green laser with already available green laser.

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years of age
* Eyes with proliferative diabetic retinopathy requiring laser photocoagulation

Exclusion Criteria:

* Eyes with media opacities not allowing proper fundus photography or adequate laser photocoagulation
* Patients requiring more than two sessions of laser photocoagulation
* Patients who had undergone previous laser photocoagulation
* Patients who had undergone any previous vitreo-retinal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-12; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Pigmentation of burn | 2 months, 4 months, 6 months post laser
Lateral spread of burn | 2 months, 4 months, 6 months post laser
Regression of new vessels | 2 months, 4 months, 6 months post laser

SECONDARY OUTCOMES:
Choroidal detachment | 2 months, 4 months, 6 months post laser
Retinal detachment | 2 months, 4 months, 6 months post laser
Tractional retinal detachment | 2 months, 4 months, 6 months post laser
Bruch's membrane rupture | 2 months, 4 months, 6 months post laser

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Mohan, MS, Principal Investigator — Arvind Eye Hospital, Madurai; Dhananjay Shukla, MS, Principal Investigator — Aravind Eye Hospital; Naresh Babu, MS, FNB, Principal Investigator — Aravind Eye Hospital
Locations (1):
- Arvind Eye Hospital, Madurai, Tamil Nadu, India